CLINICAL TRIAL: NCT04785716
Title: Real-life Use of Niraparib in a Patient Access Program in Norway
Status: Completed | Type: Observational
Sponsor: Kristina Lindemann (Other)
Collaborators: University Hospital of North Norway (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor-Investigator, Kristina Lindemann, Associate Prof. Kristina Lindemann, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Other Study IDs: REK 62008
Record Dates: First submitted 2021-01-27; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer; Peritoneal Cancer
Keywords: Poly(ADP-ribose) Polymerase Inhibitors; real life data; ovarian cancer; niraparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Niraparib — Niraparib provided through the patient access program

SUMMARY:
Retrospective observational study of patients treated with niraparib in an individual patient access program in Norway.

DETAILED DESCRIPTION:
Poly (ADP-ribose) polymerase (PARP) inhibitors have emerged as new treatment options in ovarian cancer. While there is now also evidence for the efficacy in the first line setting, they were initially studied in recurrent disease both as maintenance after chemotherapy but also as treatment on its own. The NOVA study was conducted in the maintenance setting of patients with recurrent high-grade serous ovarian-, tube or peritoneal cancer who had responded to platinum-based chemotherapy. In 2017 Tesaro opened an individual patient access program in Norway, and in July 2017 the first Norwegian patient was enrolled. We performed a retrospective observational study of patients treated with niraparib in the individual patient access program in Norway. The objective of the study is to provide preliminary efficacy and safety data in a rather unselected population of non-gBRCA patients with recurrent ovarian-, tube-, or peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the individual patient access program since 2017.
* Patients who have received at least one dose of niraparib will be included.
* Patients will be identified and recruited from the following participating sites: Oslo University Hospital, Haukeland University Hospital, Stavanger University Hospital, St. Olavs Hospital, University Hospital of Northern Norway and Sørlandet sykehus.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsed ovarian, fallopian tube or peritoneum cancer in response to platinum based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Time to first subsequent treatment | Through study completion, an average of 15 months
  Date of start of niraparib to start date of subsequent treatment

SECONDARY OUTCOMES:
Time to progression | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18.5 months
  Date of start niraparib to date of investigator assessed progression
Time to progression assesed by CA-125 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18.5 months
  Date of start niraparib to date of 2xUNL CA-125
Type of subsequent chemotherapy if applicable | Through study completion, an average of 15 months
  Type of subsequent chemotherapy
Response to subsequent chemotherapy (investigator assessed, measured as ORR and CBR | Through study completion, an average of 15 months
  Response to subsequent chemotherapy (investigator assessed, measured as ORR and CBR
Proportion of patients with at least one grade 3 and 4 hematologic and non-hematologic toxicity | Through study completion, an average of 15 months
  Proportion of patients with at least one grade 3 and 4 hematologic and non-hematologic toxicity
Frequency of dose interruptions | Through study completion, an average of 15 months
  Frequency of dose interruptions
Frequency of dose reductions | Through study completion, an average of 15 months
  Frequency of dose reductions
Reasons for discontinuation (i.e. toxicity, progressive disease, patient preferences, other) | Through study completion, an average of 15 months
  Reasons for discontinuation (i.e. toxicity, progressive disease, patient preferences, other)
Compare progression-free survival data in groups by CA 125 at baseline (normalized vs not normalized) | Through study completion, an average of 15 months
  Compare progression-free survival data in groups by CA 125 at baseline (normalized vs not normalized)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Lindemann, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital (OUH), Oslo, Norway